CLINICAL TRIAL: NCT06000072
Title: Comparison of Tele-rehabilitation or Video-Based Core Exercises in Individuals With Axial Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Özgül Öztürk, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATADEK 2023 - 10/341
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Axial Spondyloarthritis; Telerehabilitation; Exercise
MeSH Terms: conditions — Axial Spondyloarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Telerehabilitation sessions including core exercises
  Interventions: Other: Core Exercise Program
- Video-based (Active Comparator): Core exercises by watching pre-recorded videos
  Interventions: Other: Core Exercise Program

INTERVENTIONS:
Other: Core Exercise Program — Core exercises

SUMMARY:
Exercise is a core treatment method in the management of Axial Spondyloarthritis. Clinical guidelines recommend a combination of pharmacologic and non-pharmacologic approaches to reduce disease activity and symptoms and improve physical function. The COVID-19 pandemic has accelerated the provision of healthcare services remotely and the digitalization of rehabilitation services. Telerehabilitation methods provide advantages in terms of transportation, prevention of infections that may occur due to suppression of immunity with drugs, and continuity of treatment in patients with axial spondyloarthritis. In this context, it is important to evaluate the effects of remote physiotherapy and rehabilitation delivery in chronic inflammatory rheumatic diseases. This study, which will examine the effects of telerehabilitation in the disease management processes of individuals with axial spondyloarthritis, is thought to shed light on future studies.

The aim of this study was to compare the effectiveness of telerehabilitation or pre-recorded video-based core exercise program on core endurance, disease activity and physical function in subjects with axial spondyloarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 55 years old,
* Axial Spondyloarthritis diagnosed by a rheumatologist,
* Not having any orthopedic, neurological, or mental illness that would affect exercise,
* Not using any assistive device for ambulation
* People who volunteer to participate

Exclusion Criteria:

* Pregnancy, malignancy, and recent surgery
* Presence of cardiopulmonary disease
* Patients with endoprosthesis and prosthesis
* Attending a regular exercise program (Pilates, core, or yoga etc.)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Core Endurance Tests : Trunk Flexion Test | 8 weeks
  The patient will be asked to cross his/her hands over his/her chest and positioned with the trunk in 60° flexion and knees in 90° flexion. The time in this position will be measured and recorded with a stopwatch. If there is any deterioration in the patient's position, the stopwatch will be stopped and the test will be terminated.
Core Endurance Tests : Side Plank (Side Bridge Test): | 8 weeks
  The patient will be asked to lie on his/her side on the dominant side and cross his/her foot over the other foot. The non-dominant arm will be crossed over the chest and placed over the dominant shoulder. The patient will be asked to stand on the dominant forearm and elbow. The time in this position will be measured with a cronometer and recorded. If there is any deterioration in the patient's position, the stopwatch will be stopped and the test will be terminated.
Core Endurance Tests : Modified Plank | 8 weeks
  The patient will be asked to position on his/her knees and elbows with his/her face to the floor. He/she will be fixed over his/her knees with the help of a belt and the duration of his/her stay in this position will be measured and recorded with a cornometer. If there is any deterioration in the patient's position, the stopwatch will be stopped and the test will be terminated.
Core Endurance Tests : Biering-Sorenson Test | 8 weeks
  Patients will be positioned in a prone position with their spina iliaca anterior superior to the edge of the bed. Participants will be asked to extend their upper body straight forward from the edge of the table. They will be immobilized over their knees with the help of a belt and the time they stay in this position will be measured and recorded with a cornometer. If there is any deterioration in the patient's position, the stopwatch will be stopped and the test will be terminated.

SECONDARY OUTCOMES:
Bath Ankylosing Spondylitis Functional Index (BASFI) | 8 weeks
  The questionnaire used to assess physical function in patients consists of 10 items related to activities of daily living. Each item is scored between 0-10 (0 meaning no difficulty, 10 meaning impossible).
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 8 weeks
  The BASDAI is used to measure ankylosing spondylitis disease activity. In this index, fatigue, pain due to spinal and peripheral joint involvement, local tenderness at the sites of insertion, duration and severity of morning stiffness in the last 1 week are evaluated. It consists of a total of 6 items and each item is scored between 0-10 (0 meaning no difficulty, 10 meaning impossible).
Bath Ankylosing Spondylitis Metrology Index (BASMI) | 8 weeks
  It is an index that includes several measurements used to evaluate spinal mobility. These measurements are tragus-wall distance, lumbar lateral flexion test, Modified Schober test, intermalleolar distance.
Global Rating of Change (GROC) | 8 weeks
  It is used to assess the patient's current health status and to calculate the difference between the initial health status.
Pain intensity (Numeric Rating Scale/NRS) | 8 weeks
  It is a scale used to determine the severity of pain. It allows the patient to describe their pain in numbers. The scale starts with the absence of pain (0) and is expressed as unbearable pain (10 or 100).
Ankylosing Spondylitis Quality of Life | 8 weeks
  The ASQoL consists of 18 questions and patients are asked to answer yes or no to each question. The total score ranges from 0-18. Higher scores indicate a poorer quality of life.
Timed Up and Go Test | 8 weeks
  The patients sit on a chair and are asked to stand up and walk for 3 meters then sit again. The time to complete this task is recorded.
30 Seconds Sit and Stand Test | 8 weeks
  The patient sits and stands for 30 s in a chair whose height is adjusted so that the knees are 90° when seated. The number of times the patient can sit and stand during this time will be calculated and recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Haydarpasa Numune Research and Training Hospital, Istanbul
  - Acıbadem Mehmet Ali Aydınlar University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sen EN, Saritas F, Ozturk O. Synchronous and asynchronous remote core stability exercises in patients with axial spondyloarthritis: a randomized-controlled clinical trial. Ir J Med Sci. 2025 Feb;194(1):137-146. doi: 10.1007/s11845-024-03846-8. Epub 2024 Nov 26. PMID 39589722